CLINICAL TRIAL: NCT06451991
Title: The Effect of Concept Map Use in Nursing Practice on Clinical Decision Making and Reflective Thinking Levels: A Randomized Controlled Study
Brief Title: The Effect of Concept Map Use in Nursing Practice
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nilgun Sert Bas (Other)
Responsible Party: Sponsor-Investigator, Nilgun Sert Bas, Lecturer, Ankara Medipol University
Organization: Ankara Medipol University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: E-81477236-604.01.01-2747
Record Dates: First submitted 2024-06-05; First posted 2024-06-11 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2024-07

CONDITIONS: Student; Educational Problems
Keywords: Nursing education; Concept map; Reflective thinking; Clinical decision making

STUDY DESIGN:
Masking Description: Within the scope of the research, students will be divided into control (n=33) and experimental (n=33) groups by simple randomisation method. Since the students and instructors should know and follow the material to be used in the data collection process, blinding was not performed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Traditional (No Intervention): The control group will use the traditional method data collection form and care plan.
- Concept Map (Experimental): The experimental group will collect data and make a maintenance plan by using a concept map after the training.
  Interventions: Other: Use of concept map in clinical practice in nursing students

INTERVENTIONS:
Other: Use of concept map in clinical practice in nursing students — Concept map will be used in clinical practice in nursing students.
  Arms: Concept Map

SUMMARY:
The aim of this randomised controlled trial is to evaluate the effect of data collection and creating a patient care plan using a concept map on the student s clinical decision-making and reflective thinking skills of students taking the surgical diseases nursing course who are in the hospital for clinical practice.

DETAILED DESCRIPTION:
With the rapid development and change in technology and modern medicine, expectations, tendencies, personality characteristics and learning styles of individuals change. At the same time, today s modern medical environment requires nurses to have analytical thinking, independent decision-making and application skills in clinical practice. One of the main objectives of nursing education is to provide students with critical thinking and decision-making skills and to reflect what they have learnt in theory to their clinical practice skills. The World Health Organisation also recommends the use of innovative and active learning methods, appropriate teaching materials and learning techniques in nursing education. One of the most important modern teaching methods that will facilitate meaningful learning among students is concept maps developed on the basis of Ausubel s Learning Assimilation Theory. At the same time, clinical decision making and reflective thinking are important elements in nursing practice and undergraduate nursing education. One of the most important goals of nursing education is to provide educational approaches to develop these concepts.

The main question[s] it aims to answer are:

* Does collecting data from the patient using a concept map instead of a traditional care plan in the clinic affect student s; clinical decision-making level?
* Does preparing a patient care plan using a concept map instead of a traditional care plan in the clinic affect student s; reflective thinking skill level in the clinic?

Research Process:

* Both groups will be administered sociodemographic data form, clinical decision-making scale in nursing, reflective thinking determination scale and teaching material evaluation form as face-to-face pre-test before the training.
* The control group will use the traditional method data collection form and care plan.
* The experimental group will be given face-to-face training before starting the application. The scope of the training will consist of the definition of concept mapping, the aims and benefits of its use in the nursing education process, the principles of concept mapping, the introduction of the materials to be used in the process of data collection and care plan preparation, concept mapping examples specific to 3 different medical cases to improve nursing student s; understanding and comprehension of concept mapping and to increase their interest in learning techniques.
* After the training, students will be asked to collect data and make a care plan using a concept map.
* After data collection, face-to-face sociodemographic data form, clinical decision-making scale in nursing, scale for determining the level of reflective thinking and teaching material evaluation form will be applied as a post-test. Population and sample: G*Power 3.1.9.7 sampling calculation programme was used to calculate the sample size in the study. Considering the mean±standard deviation values of the Clinical Decision Making in Nursing scale, the total sample size was calculated as 56, with a minimum of 28 for each group, with an effect size of 0.79 and a margin of error of ± 0.05 at the 82% confidence interval level. However, the research will be started with 33 participants by taking 20% more than the sample size determined by taking into account the situation of the participants leaving the research during the process.

Statistical Method(s): The data obtained from the study will be evaluated using Statistical Package for the Social Sciences (SPSS) for Windows version 25.0 programme. Number, percentage, standard deviation, mean, min-max values will be used to define the data. According to the measurement level of the data, correlation analysis or chi-square dependency tests will be used for the relationships between variables. The suitability of continuous variables for normal distribution will be evaluated by Kolmogrov-Simirnov test. In group comparisons, Anova will be used for variables that fit the normal distribution, Kruskal Wallis and Mann Whitney U tests will be used for variables that do not fit the normal distribution. 0,05 will be used as significance level, and it will be stated that there is a significant difference in case of ia small 0,05, and there is no significant difference in case of is small 0,05.

The researchers will compare the control and experimental groups to see whether the use of concept maps in clinical practice has an effect on student s; clinical decision-making and reflective thinking skills.

It is thought that the data obtained as a result of the study will support innovative applications, and at the same time, it will be explanatory and guiding about whether the use of concept maps is effective in developing student s; clinical decision-making and reflective thinking skills.

ELIGIBILITY:
Inclusion Criteria:

* To be taking surgical diseases nursing course
* To agree to participate in the study

Exclusion Criteria:

* To have received training on concept mapping before the study
* Not participating in the training given by the researchers before the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2025-03-03 (Actual); Primary Completion 2025-05-13 (Actual); Study Completion 2025-05-13 (Actual)

PRIMARY OUTCOMES:
Clinical Decision Making Scale in Nursing | 3 weeks
  The scale consists of 40 items. The scale includes four sub-dimensions (10 items each), namely "investigating options and ideas", "investigating goals and values", "evaluating results" and "investigating knowledge and adopting new knowledge impartially". The scale is 5-point Likert type. The minimum total score of the scale is 40 points and the maximum score is 200 points. Cronbach Alpha reliability coefficient is 0.78.
Determination of Reflective Thinking Scale | 3 weeks
  The scale is 5-point Likert type and consists of 16 items. The scale measures students' reflective thinking skill levels at the end of a lesson in four sub-dimensions, each consisting of four items: habit, comprehension, reflection and critical reflection. The lowest score that can be obtained from each sub-dimension is 4 and the highest score is 20. Cronbach Alpha reliability coefficient is 0.77.

SECONDARY OUTCOMES:
Teaching Material Evaluation Form | 3 weeks
  This form was created by the researchers for the evaluation of the teaching material used. The form consists of 16 items evaluating its effect on clinical practice such as its effect on satisfaction, effect on motivation, effect on critical thinking, effect on problem solving skills, effect on holistic approach, effect on learning. Visual analogue scale (VAS) was used to evaluate these items. The VAS was modified by rephrasing the original scale to assess and measure the traditional or concept map data collection and patient care plan form used by the students. The VAS consists of a straight line from zero to 100. It will be measured and evaluated by the researchers after the students' marking.

CONTACTS AND LOCATIONS:
Overall Officials: Nilgün Sert Baş, RN, MSc, Principal Investigator — Ankara Medipol University
Locations (1):
- Ankara Medipol University, Ankara, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Culha, I. Active learning methods used in nursing education. Journal of Pedagogical Research, 2019; 3(2), 74-86.
- [Background] Wu HZ, Wu QT. Impact of mind mapping on the critical thinking ability of clinical nursing students and teaching application. J Int Med Res. 2020 Mar;48(3):300060519893225. doi: 10.1177/0300060519893225. PMID 32212879
- [Background] World Health Organization.
- [Background] Amaniyan S, Pouyesh V, Bashiri Y, Snelgrove S, Vaismoradi M. Comparison of the Conceptual Map and Traditional Lecture Methods on Students' Learning Based on the VARK Learning Style Model: A Randomized Controlled Trial. SAGE Open Nurs. 2020 Jul 8;6:2377960820940550. doi: 10.1177/2377960820940550. eCollection 2020 Jan-Dec. PMID 33415293
- [Background] Tutticci N, Lewis PA, Coyer F. Measuring third year undergraduate nursing students' reflective thinking skills and critical reflection self-efficacy following high fidelity simulation: A pilot study. Nurse Educ Pract. 2016 May;18:52-9. doi: 10.1016/j.nepr.2016.03.001. Epub 2016 Mar 15. PMID 27235566
- [Background] Karacabay, K, Savcı A, Öztürk B. Cerrahi Hastalıkları Hemşireliği Dersi Alan Öğrencilerin Kendi Kendine Öğrenme, Klinik Karar Verme ve Yansıtıcı Düşünme Düzeylerinin İncelenmesi. İnönü Üniversitesi Sağlık Hizmetleri Meslek Yüksek Okulu Dergisi 10.2 (2022): 667-680.